CLINICAL TRIAL: NCT04196127
Title: Bite Force and Muscle Function in Patients With Tension-type Headache
Brief Title: Jaw Muscle Function in Patients With Tension-type Headache
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Danish Headache Center (Other)
Collaborators: UMC Utrecht (Other); Academic Centre for Dentistry in Amsterdam (Other)
Responsible Party: Principal Investigator, Bjarne Kjeldgaard Madsen, Physiotherapist, PhD, Danish Headache Center
Other Study IDs: 091219
Record Dates: First submitted 2019-12-06; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Headache Disorders; Tension-Type Headache
Keywords: Bite force; Temporomandibular disorder; Neck pain
MeSH Terms: conditions — Headache Disorders; Tension-Type Headache; Temporomandibular Joint Disorders; Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TTH: Patients with tension-type headache. They may not experience migraine, but can experience neck pain and/or temporomandibular dysfunction.
  Interventions: Other: Bite force testing
- Healthy controls: Participants without frequent headaches. They may experience neck pain and/or temporomandibular dysfunction.
  Interventions: Other: Bite force testing

INTERVENTIONS:
Other: Bite force testing — Maximum bite force examination with a force intra-oral measuring device

SUMMARY:
Patients with tension-type headache (TTH) and migraine often experience musculoskeletal complaints, like neck pain and/or jaw pain. Earlier studies have revealed an association between different headache types and neck pain and discussed the possible role of the cervical muscles. Furthermore, patients with neck pain show a decrease in motor control of the jaw, without having any other signs of TMD. Similarly, studies in patients with TMD have only found an indication for poorer neck muscle function. Patients with TMD also show a decrease in bite force and force steadiness compared to healthy controls. It is however, unknown if bite force and force steadiness are similarly impaired in patients with headache and/or neck pain.

The current study will take a closer look at the jaw muscle function of in patients with TTH, with and without neck pain.

DETAILED DESCRIPTION:
Tension-type headache (TTH) and migraine has been found to coincide with cervical pain, musculoskeletal dysfunction and/or temporomandibular disorders (TMD). The possible interplay between these three symptoms/disorders, headache, neck pain and TMD, have not been studied completely, only in sections. Earlier studies have revealed an association between different headache types and neck pain and discussed the possible role of the cervical muscles. Patients with TTH and (chronic) migraine exhibit lower muscle strength in the neck extensor muscles compared to healthy controls. Patients with neck pain show a decrease in motor control of the jaw, without having any other signs of TMD. Similarly, studies in patients with TMD have only found an indication for poorer neck muscle function while patients with TMD also show a decrease in bite force and force steadiness compared to healthy controls. It is however, unknown if bite force and force steadiness are similarly impaired in patients with headache and/or neck pain.

Muscle tenderness increases with increasing headache frequency and intensity in TTH while this association is not present in migraine patients. Tenderness has a significant influence on the neck muscle function in TTH patients and there is a negative correlation between Total Tenderness (TTS) and muscle force. There is currently, however, no clear understanding of the influence of tenderness on the function of jaw muscles in TTH patients.

The current project will increase the investigator's understanding of the interplay or dependency between the function of the jaw and neck muscles in TTH patients. If a comorbidity of TMD or neck pain make TTH patients more prone to dysfunction of jaw and neck muscles, this may lead to a subgrouping of these TTH patients. Together with the muscle function deficits discovered in the current case control study, this may suggest a targeted treatment for TTH to be tested in a follow up randomized control study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 55 years old.
* Diagnosed Frequent episodic TTH (1-14 headache days / month) or chronic TTH (≥15 headache days/ month) based on the ICHD-3.
* Maximum 3 days of migraine per month.
* Signed informed acceptance of participation.

Exclusion Criteria:

* medication overuse headache (ICHD-3)
* missing more than 1 molar,
* previous whiplash or head trauma,
* other major physical or neurological diseases,
* diagnosed depression, other mental illness
* unable to understand and speak Danish.
* Pregnant or lactating women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be recruited from the Danish Headache Center. Additionally the patients and healthy controls will be included from a Danish web page for trials www.forsoegsperson.dk and from a research data base in Danish Headache Center during 2019-2020. When the participants respond through the webpage through either mail or telephone, they will receive written information through mail. They will be informed that they have the right to take a family member or close related, And that the oral information will be postponed till all can participate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-06 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Bite Force | baseline
  Maximum bite force in Newton, best out of three tests

SECONDARY OUTCOMES:
Bite Force Steadiness | baseline
  30% of maximum bite force held for 30 seconds, expressed as mean and standard deviation
Neck muscle function | baseline
  Ratio of flexion/extension strength
Total Tenderness Score | baseline
  Overall total tenderness score (range 0 - 48; higher score means higher tenderness of the muscles).
Total Tenderness Score | Immediately after muscle function testing (outcomes 1-3)
  Overall total tenderness score (range 0 - 48; higher score means higher tenderness of the muscles).

OTHER OUTCOMES:
Numeric Pain Rating Scale | baseline
  Pain intensity for headache, neck pain and jaw complaints (range 0 - 10; higher means more pain)
Numeric Pain Rating Scale | Immediately after muscle function testing (outcomes 1-3)
  Pain intensity for headache, neck pain and jaw complaints (range 0 - 10; higher means more pain)
Prevalence of temporomandibular disorders | baseline
  The prevalence of the different diagnoses of temporomandibular disorders, based on the diagnostic criteria for temporomandibular disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Bjarne Kjeldgaard Madsen, PT, PhD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center Rigshospitalet - Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Armijo-Olivo S, Warren S, Fuentes J, Magee DJ. Clinical relevance vs. statistical significance: Using neck outcomes in patients with temporomandibular disorders as an example. Man Ther. 2011 Dec;16(6):563-72. doi: 10.1016/j.math.2011.05.006. Epub 2011 Jun 12. PMID 21658987
- [Background] Ashina S, Bendtsen L, Lyngberg AC, Lipton RB, Hajiyeva N, Jensen R. Prevalence of neck pain in migraine and tension-type headache: a population study. Cephalalgia. 2015 Mar;35(3):211-9. doi: 10.1177/0333102414535110. Epub 2014 May 22. PMID 24853166
- [Background] Ballenberger N, von Piekartz H, Danzeisen M, Hall T. Patterns of cervical and masticatory impairment in subgroups of people with temporomandibular disorders-an explorative approach based on factor analysis. Cranio. 2018 Mar;36(2):74-84. doi: 10.1080/08869634.2017.1297904. Epub 2017 Mar 20. PMID 28317439
- [Background] Bendtsen L, Fernandez-de-la-Penas C. The role of muscles in tension-type headache. Curr Pain Headache Rep. 2011 Dec;15(6):451-8. doi: 10.1007/s11916-011-0216-0. PMID 21735049
- [Background] Fernandez-de-las-Penas C, Perez-de-Heredia M, Molero-Sanchez A, Miangolarra-Page JC. Performance of the craniocervical flexion test, forward head posture, and headache clinical parameters in patients with chronic tension-type headache: a pilot study. J Orthop Sports Phys Ther. 2007 Feb;37(2):33-9. doi: 10.2519/jospt.2007.2401. PMID 17366957
- [Background] Florencio LL, de Oliveira AS, Carvalho GF, Tolentino Gde A, Dach F, Bigal ME, Fernandez-de-las-Penas C, Bevilaqua Grossi D. Cervical Muscle Strength and Muscle Coactivation During Isometric Contractions in Patients With Migraine: A Cross-Sectional Study. Headache. 2015 Nov-Dec;55(10):1312-22. doi: 10.1111/head.12644. Epub 2015 Sep 21. PMID 26388193
- [Background] de Groot RJ, Wetzels JW, Merkx MAW, Rosenberg AJWP, de Haan AFJ, van der Bilt A, Abbink JH, Speksnijder CM. Masticatory function and related factors after oral oncological treatment: A 5-year prospective study. Head Neck. 2019 Jan;41(1):216-224. doi: 10.1002/hed.25445. Epub 2018 Dec 15. PMID 30552819
- [Background] Madsen BK, Sogaard K, Andersen LL, Skotte JH, Jensen RH. Neck and shoulder muscle strength in patients with tension-type headache: A case-control study. Cephalalgia. 2016 Jan;36(1):29-36. doi: 10.1177/0333102415576726. Epub 2015 Apr 1. PMID 25834271
- [Background] Madsen BK, Sogaard K, Andersen LL, Skotte J, Tornoe B, Jensen RH. Neck/shoulder function in tension-type headache patients and the effect of strength training. J Pain Res. 2018 Feb 23;11:445-454. doi: 10.2147/JPR.S146050. eCollection 2018. PMID 29503581
- [Background] Testa M, Geri T, Gizzi L, Petzke F, Falla D. Alterations in Masticatory Muscle Activation in People with Persistent Neck Pain Despite the Absence of Orofacial Pain or Temporomandibular Disorders. J Oral Facial Pain Headache. 2015 Fall;29(4):340-8. doi: 10.11607/ofph.1432. PMID 26485381
- [Background] Testa M, Geri T, Pitance L, Lentz P, Gizzi L, Erlenwein J, Petkze F, Falla D. Alterations in jaw clenching force control in people with myogenic temporomandibular disorders. J Electromyogr Kinesiol. 2018 Dec;43:111-117. doi: 10.1016/j.jelekin.2018.07.007. Epub 2018 Jul 26. PMID 30269020
- [Background] van der Meer HA, Speksnijder CM, Engelbert RHH, Lobbezoo F, Nijhuis-van der Sanden MWG, Visscher CM. The Association Between Headaches and Temporomandibular Disorders is Confounded by Bruxism and Somatic Symptoms. Clin J Pain. 2017 Sep;33(9):835-843. doi: 10.1097/AJP.0000000000000470. PMID 28002094
- [Background] von Piekartz H, Pudelko A, Danzeisen M, Hall T, Ballenberger N. Do subjects with acute/subacute temporomandibular disorder have associated cervical impairments: A cross-sectional study. Man Ther. 2016 Dec;26:208-215. doi: 10.1016/j.math.2016.09.001. Epub 2016 Sep 23. PMID 27744136